CLINICAL TRIAL: NCT05303792
Title: A Randomized Phase II Study Comparing Inotuzumab Plus Chemotherapy Versus Standard Chemotherapy in Older Adults With Philadelphia-Chromosome-Negative B-Cell Acute Lymphoblastic Leukemia
Brief Title: Testing the Combination of Inotuzumab Ozogamicin and Lower Dose Chemotherapy Compared to Usual Chemotherapy for Adults With B-Cell Acute Lymphoblastic Leukemia or B-Cell Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A042001; NCI-2022-01735 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Vincristine; Dexamethasone; Inotuzumab Ozogamicin; Methotrexate; Cytarabine; Methylprednisolone; Rituximab; Prednisone; Mercaptopurine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (inotuzumab ozogamicin, chemotherapy) (Experimental): Induction: For cycles 1-4 on days 2 and 8, patients receive inotuzumab ozogamicin IV and IT chemotherapy consisting of alternating Cytarabine and Methotrexate. Patients with leukemic blasts expressing CD20 also receive rituximab IV on days 2 and 8 of cycles 1-4. For cycles 1,3,5,7, patients receive cyclophosphamide intravenously (IV) on days 1-3, mesna IV, vincristine IV on days 1 and 8, and dexamethasone IV or orally (PO) on days 1-4 and 11-14. For cycles 2,4,6,8, patients receive methotrexate on day 1, cytarabine IV on days 2-3, and methylprednisolone on days 1-3. Patients >= 70 years of age receive either 2 or 4 cycles of treatment. Patients < 70 years of age receive up to 8 cycles of treatment.
  Maintenance: Patients receive vincristine IV on day 1, prednisone PO on days 1-5, mercaptopurine PO on days 1-28, and methotrexate PO weekly. Treatment occurs for up to 24 cycles or 2 years, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Dexamethasone; Biological: Inotuzumab Ozogamicin; Drug: Methotrexate; Drug: Cytarabine; Drug: Methylprednisolone; Biological: Rituximab; Drug: Prednisone; Drug: Mercaptopurine
- Arm B (chemotherapy) (Active Comparator): Induction: For cycles 1-4 on days 2 and 8, patients receive IT chemotherapy consisting of alternating Cytarabine and Methotrexate. Patients with leukemic blasts expressing CD20 also receive rituximab IV on days 2 and 8 of cycles 1-4. For cycles 1,3,5,7, patients receive cyclophosphamide intravenously (IV) on days 1-3, mesna IV, doxorubicin IV on day 4, vincristine IV on days 1 and 8, and dexamethasone IV or orally (PO) on days 1-4 and 11-14. For cycles 2,4,6,8, patients receive methotrexate on day 1, cytarabine IV on days 2-3, and methylprednisolone on days 1-3. Patients >= 70 years of age receive either 2 or 4 cycles of treatment. Patients < 70 years of age receive up to 8 cycles of treatment.
  Maintenance: Patients receive vincristine IV on day 1, prednisone PO on days 1-5, mercaptopurine PO on days 1-28, and methotrexate PO weekly. Treatment occurs for up to 24 cycles or 2 years, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine; Drug: Methylprednisolone; Biological: Rituximab; Drug: Prednisone; Drug: Mercaptopurine; Drug: Doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
Drug: Vincristine — Given IV
Drug: Dexamethasone — Given IV or PO
Biological: Inotuzumab Ozogamicin — Given IV
  Arms: Arm A (inotuzumab ozogamicin, chemotherapy)
Drug: Methotrexate — Given IV or PO
Drug: Cytarabine — Given IV
Drug: Methylprednisolone — Given IV
Biological: Rituximab — Given IV
Drug: Prednisone — Given PO
Drug: Mercaptopurine — Given PO
Drug: Doxorubicin — Given IV
  Arms: Arm B (chemotherapy)

SUMMARY:
This phase II trial compares the combination of inotuzumab ozogamicin and chemotherapy to the usual chemotherapy in treating patients with B-cell acute lymphoblastic leukemia or B-cell lymphoblastic lymphoma. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a drug, called CalichDMH. Inotuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD22 receptors, and delivers CalichDMH to kill them. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving inotuzumab ozogamicin with chemotherapy may help shrink the cancer and stop it from returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare undetectable measurable residual disease (MRD) event-free survival (EFS) rate of the experimental arm (A) to standard arm (B) with EFS defined as time from randomization to occurrence of an event.

SECONDARY OBJECTIVES:

I. To determine overall response rate (complete response [CR], CR + complete remission with incomplete platelet counts [CRp], CR + complete remission with partial hematologic recovery [CRh], CR + complete remission with incomplete blood count recovery [CRi]) at designated time points (after cycle 1, after cycle 2, end of intensive phase) in each treatment arm.

II. To determine rate of flow cytometry MRD-negativity (undetectable or detectable < 10^-4) at designated time points (after cycle 1, after cycle 2, end of intensive phase) in each treatment arm.

III. To compare MRD response by central aspirate multiparameter flow cytometry (Wood lab) to next generation sequencing MRD assessment (clonoSEQ, Adaptive) of blood and bone marrow at designated time points (after cycle 1, after cycle 2, and end of intensive phase) and to determine association with outcome, in each treatment arm.

IV. To determine the event-free survival (EFS) standard-definition (event defined as failure to achieve morphologic remission by cycle 2, hematologic relapse, death), disease-free survival (DFS), overall survival (OS) of each arm (median, 6-month, 1-year, 2-year, 3-year) in each treatment arm.

V. To determine proportion of patients who proceed to allogeneic transplant after initial response (without intervening salvage therapy) in each treatment arm.

VI. To determine rate of liver toxicity (grade 3-5 alanine aminotransferase [ALT] increase, aspartate aminotransferase [AST] increase, bilirubin increase, alkaline phosphatase increase).

VII. To describe the safety and tolerability of each arm including rate of grade 3-5 non-hematologic toxicity and treatment-related mortality (grade 5 toxicity VIII. To determine rate of delays in intensive-phase chemotherapy due to neutropenia and thrombocytopenia (in responding patients).

IX. To assess the baseline variations in comorbidity burden, physical, nutritional, and cognitive function of the study participants, and explore the association between comorbidity burden, physical, nutritional, and cognitive function, and the outcomes of therapy (grade 3-5 non-hematological toxicities, and OS).

X. To explore the longitudinal changes in physical, nutritional, and cognitive function among the experimental and control groups.

XI. To compare the burden of patient-reported symptomatic adverse events between treatment arms using the Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE).

XII. To correlate specific karyotype groups (normal or various primary and secondary chromosomal abnormalities) with clinical and laboratory parameters.

XIII. To correlate specific karyotype groups with response rates, response duration, MRD, and survival in patients treated on this study.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

INDUCTION: Patients receive cyclophosphamide intravenously (IV) over 3 hours every 12 hours (Q12H) on days 1-3 of cycles 1, 3, 5, and 7, vincristine IV on days 1 and 8 of cycle 1, 3, 5, and 7, dexamethasone IV or orally (PO) on days 1-4 and 11-14 of cycles 1, 3, 5, and 7, inotuzumab ozogamicin IV over 1 hour on days 2 and 8 of cycles 1-4, methotrexate IV over 24 hours on day 1 of cycles 2, 4, 6, and 8, cytarabine IV over 3 hours Q12H on days 2-3 of cycles 2, 4, 6, and 8, and methylprednisolone IV over 2 hours Q12H on days 1-3. Patients with leukemic blasts expressing CD20 also receive rituximab IV on days 2 and 8 of cycles 1-4. For patients >= 70 years of age, treatment repeats every 28 days for 2 cycles (an additional 2 cycles may be given at the discretion of the principal investigator [PI]) in the absence of disease progression or unacceptable toxicity. For patients < 70 years of age, treatment repeats every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on day 1, prednisone PO daily on days 1-5, mercaptopurine PO twice daily (BID) on days 1-28, and methotrexate PO weekly. Treatment repeats every 28 days for up to 24 cycles or 2 years, whichever comes first, in the absence of disease progression or unacceptable toxicity.

ARM B:

INDUCTION: Patients receive cyclophosphamide IV over 3 hours Q12H on days 1-3 of cycle 1, 3, 5, and 7, vincristine IV on days 1 and 8 of cycles 1, 3, 5, and 7, dexamethasone IV or PO on days 1-4 and 11-14 of cycle 1, 3, 5, and 7, doxorubicin IV over 24 hours on day 4 of cycles 1, 3, 5, and 7, methotrexate IV over 24 hours on day 1 of cycles 2, 4, 6, and 8, cytarabine IV over 3 hours Q12H on days 2-3 of cycles 2, 4, 6, and 8, and methylprednisolone IV over 2 hours Q12H on days 1-3 of cycles 2, 4, 6, and 8. Patients with leukemic blasts expressing CD20 also receive rituximab IV on days 2 and 8 of cycles 1-4. For patients >= 70 years of age, treatment repeats every 28 days for 2 cycles (an additional 2 cycles may be given at the discretion of the PI) in absence of disease progression or unacceptable toxicity. For patients < 70 years of age, treatment repeats every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on day 1, prednisone PO daily on days 1-5, mercaptopurine PO BID on days 1-28, and methotrexate PO weekly. Treatment repeats every 28 days for up to 24 cycles or 2 years, whichever comes first, in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months until 1 year after completion of therapy, every 3 months until 2 years after completion of therapy, and then every 6 months until 5 years from study registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA (STEP 0)
* Research bone marrow or peripheral blood submission

  * This bone marrow or peripheral blood submission is mandatory prior to registration/randomization as baseline for real-time MRD analysis. The bone marrow sample should be from the first aspiration (i.e., first pull). Aspirate needle should be redirected if needed to get first pull bone marrow aspirate. It should be obtained as soon after pre-registration as possible
* REGISTRATION INCLUSION CRITERIA (STEP 1)
* Diagnosis of B-cell acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LBL) per World Health Organization (WHO) 2016 criteria. Patients must have >= 5% blasts in the bone marrow or blood. Patients with lymphoblastic lymphoma (LBL) without measurable marrow involvement (>= 5% blasts) are not eligible

  * T-cell ALL/LBL, Philadelphia-chromosome positive B-cell (as determined by fluorescence in situ hybridization [FISH], cytogenetics, or reverse transcriptase polymerase chain reaction [RT-PCR]), and Burkitt's like leukemia/lymphoma (mature B-ALL) are not eligible
* Must be CD22 positive by local assessment (>= 20% by immunohistochemistry or flow cytometry). Patients are eligible regardless of CD20 status but CD20 expression should be assessed at diagnosis by flow cytometry or immunohistochemistry
* Patients must have >= 5% blasts in the bone marrow or blood. Patients with lymphoblastic lymphoma (LBL) without marrow involvement (>= 5% blasts) are not eligible
* No prior chemotherapy for ALL except for hydroxyurea (no limit), steroids limited to 7 days, ATRA (no limit), vincristine (single dose), and/or intra-thecal chemotherapy. Leukapheresis is permitted. Palliative radiation to doses 24 Gy or less is permitted. Patients being treated with chronic steroids for other reasons (autoimmune disorder, etc.) are eligible
* Age >= 50 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2. ECOG 3 permitted if related to disease
* Creatinine =< 2.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * Except in the event of: 1) Gilbert disease, in which case total bilirubin must be =< 2 x ULN, or 2) elevated bilirubin believed by investigator to be due to leukemic infiltration, in which case total bilirubin must be =< 2 x ULN
* AST / ALT =< 2.5 x upper limit of normal (ULN)
* Cardiac ejection fraction (as measured by multigated acquisition scan [MUGA] or echocardiogram) > 40%
* No clinically relevant liver disease (such as cirrhosis, active hepatitis, or alcohol use disorder), which in the opinion of the treating physician would make this protocol unreasonably hazardous

  * Patients with known hepatitis B virus (HBV) infection are eligible if they are on effective HBV suppressive therapy with undetectable HBV viral load and there is no clinically relevant liver disease present (related or unrelated to HBV-related liver damage)
  * Patients with known history of hepatitis C virus (HCV) infection are eligible if they have cleared the infection spontaneously or via eradication therapy (HCV viral load undetectable) and there is no clinically relevant liver disease present (related or unrelated to HCV-related liver damage)
* Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Include as applicable: Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom)

Exclusion Criteria:

* Physicians should consider whether any of the following may render the patient inappropriate for this protocol:

  * Medical condition such as uncontrolled diabetes mellitus, uncontrolled cardiac disease, and uncontrolled pulmonary disease.
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * Patients with a "currently active" second malignancy other than non-melanoma skin cancers, early stage prostate cancer, cervical carcinoma in situ, or other cancer for which standard of care would be observation (not requiring treatment). Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 1 year, or if the cancer has been surgically resected and considered cured. Patients with a history of multiple myeloma with absence of serum paraprotein for >= 1 year are not considered to have a "currently active" malignancy.
* REGISTRATION EXCLUSION CRITERIA (STEP 1)
* Patients with symptomatic central nervous system (CNS) disease are not eligible. CNS assessment is not required for eligibility determination if asymptomatic

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | From randomization to failure to achieve measurable residual disease (MRD)-negative complete response (CR) after two cycles of chemotherapy, relapse, or death from any causes, assessed at 2 months (after 2 cycles of treatment)
  Will be evaluated using the methods of Kaplan-Meier as well as Cox regression models.

SECONDARY OUTCOMES:
Disease-free survival | Time from achieving a CR/ complete remission with incomplete blood count recovery (CRi) to the time of relapse and/or death, assessed up to 5 years
  Will be evaluated using the methods of Kaplan-Meier as well as Cox regression models.
Overall survival | From randomization to the time of death due to any cause, assessed up to 5 years
  Will be evaluated using the methods of Kaplan-Meier as well as Cox regression models.
Complete remission rate | Up to 5 years
  The proportion of patients who achieve complete remission or any response to induction therapy will be summarized as the proportion of patients who achieve any type of response to induction therapy divided by the number of all evaluable patients registered to this trial and who received at least one dose of induction therapy. Corresponding 95% binomial confidence intervals will also be calculated. In a similar manner, the investigators will also evaluate the overall induction response rates. All evaluable patients will be used for this analysis.
Overall response rate | Up to 5 years
  Overall response rate (CR/CRi, CR/complete remission with incomplete platelet counts [CRp], CR/complete remission with partial hematologic recovery [CRh]). The proportion of patients who achieve complete remission or any response to induction therapy will be summarized as the proportion of patients who achieve any type of response to induction therapy divided by the number of all evaluable patients registered to this trial and who received at least one dose of induction therapy. Corresponding 95% binomial confidence intervals will also be calculated. In a similar manner, the investigators will also evaluate the overall induction response rates. All evaluable patients will be used for this analysis.
MRD-negativity rate | Up to end of cycle 8 (1 cycle = 28 days)
  MRD-negativity by flow cytometry will be evaluated at designated time point (after cycle 1, after cycle 2, end of intensive phase). Will also compare MRD assessment by centralized aspirate flow cytometry (Wood lab) to next generation sequencing (clonoSEQ, Adaptive) of blood and bone marrow at designated time points; and determine association with outcome.
Event-free survival | Up to 5 years
  Event defined as failure to achieve Complete Response (CR)/Complete Remission with Incomplete Blood Count Recovery (CRi)/Complete Remission with Partial Hematological Recovery (CRh)/Complete Remission with Incomplete Platelet Counts (CRp), relapse, death.
Rate of grade 3-5 adverse events | Up to 5 years
  The proportion of patients experiencing a grade 3+ adverse events or toxicities will be described for each treatment arm, but will also be compared between the arms using Fisher's exact tests.

CONTACTS AND LOCATIONS:
Overall Officials: Marlise R. Luskin, MD, MSCE, Study Chair — Dana-Farber Cancer Institute
Locations (72):
- United States (71):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- San Juan City Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided